CLINICAL TRIAL: NCT01093716
Title: Comparison of Anti-craving Efficacy of Right and Left Prefrontal High Frequency rTMS in Alcohol Dependence: a Randomized Double-blind Study
Brief Title: Anti-craving Efficacy of Right and Left Prefrontal High Frequency Repetitive Transcranial Magnetic Stimulation (rTMS) in Alcohol Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Psychiatry, Ranchi, India (Other)
Responsible Party: Prof. S. Haque Nizamie, Central Institute of Psychiatry, Ranchi, India
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADSTMS2010
Record Dates: First submitted 2010-03-22; First posted 2010-03-26 (Estimated); Last update posted 2010-03-26 (Estimated); Status verified 2010-03

CONDITIONS: Alcohol Dependence
Keywords: Alcohol dependence; Craving; rTMS; Dorsolateral prefrontal cortex
MeSH Terms: conditions — Alcoholism | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rTMS (Experimental): Compare the change in craving parameters following high frequency rTMS stimulation of right and left DLPFC in patients with alcohol dependence
  Interventions: Device: Magstim Rapid® (rTMS)

INTERVENTIONS:
Device: Magstim Rapid® (rTMS) — Ten daily sessions of rTMS treatments using Magstim Rapid® device (10 Hz, 110% of the MT, 4.9 seconds per train, inter-train interval of 30 seconds, and 20 trains per session) with an air cooled figure-of-eight coil over either right or left DLPFC

SUMMARY:
Null hypothesis: There will be no significant difference in the change in craving parameters between right and left prefrontal high frequency rTMS in patients with alcohol dependence.

DETAILED DESCRIPTION:
The patients clinically diagnosed as Alcohol dependence syndrome (F 10.24) according to ICD-10 DCR, fulfilling the inclusion and exclusion criteria will be taken up for the study. A detailed physical examination will be done to rule out any major medical or neurological disease. Written informed consent will be taken after explaining the objectives and procedure of the study in detail. To ensure that the patients selected are right handed, Handedness Preference Schedule will be applied. Socio-demographic data will be collected. Baseline SADQ-C and CIWA-Ar will be administered to determine the severity of alcohol dependence and the intensity of withdrawal symptoms respectively. When the CIWA-Ar score becomes ≤ 10, then they will be taken up for rTMS application. For these patients baseline ACQ-NOW will be administered to measure the baseline craving. Patients will be randomly allocated into two groups using randomization table. The first group will receive active rTMS of the right pre-frontal cortex; the second group will be administered active rTMS of the left pre-frontal cortex. Each patient will receive rTMS sessions 5 days a week for 2 weeks. ACQ-NOW score will again be documented in both the groups after the last rTMS session to observe the changes in craving parameters. The rating will be done by one of the authors who will be blind to the nature of rTMS stimulation being administered to the patients.

The motor threshold (MT) for the left abductor pollicis brevis will be determined by a figure of 8 shaped coil, using the Rossini-Rothwell method. MT will be defined as the lowest intensity, which produces 5 motor evoked potential (MEP) responses of at least 50 µV in 10 trials. The prefrontal cortex rTMS stimulation site will be determined by measuring 5 cm anterior and in a parasagittal line from the point of maximum stimulation of left abductor pollicis muscle. Ten active rTMS treatments will be administered at 10 Hz frequency, over right or left prefrontal cortex at 110% of MT for duration of 5 seconds and 20 trains per session, with the coil-angled tangentially to the head.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Alcohol dependence syndrome according to ICD-10 DCR,
2. Male patients aged between 18-60 years,
3. Patients with CIWA-Ar scores ≤10,
4. Right handed, normotensive patients,
5. Patients giving written informed consent.

Exclusion Criteria:

1. Comorbid psychiatric, major medical or neurological disorders,
2. History of withdrawal seizures, delirium tremens or significant head injury,
3. Subjects with pacemaker or metal in any part of the body excluding the mouth.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2009-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Craving | 2 weeks
  Alcohol Craving Questionnaire (ACQ-NOW) total score

SECONDARY OUTCOMES:
Craving | 2 weeks
  Alcohol Craving Questionnaire (ACQ-NOW) factor scores

CONTACTS AND LOCATIONS:
Overall Officials: S Haque Nizamie, Principal Investigator — Central Institute of Psychiatry, Kanke, Ranchi, Jharkhand, India

REFERENCES:
- [Derived] Mishra BR, Praharaj SK, Katshu MZ, Sarkar S, Nizamie SH. Comparison of anticraving efficacy of right and left repetitive transcranial magnetic stimulation in alcohol dependence: a randomized double-blind study. J Neuropsychiatry Clin Neurosci. 2015 Winter;27(1):e54-9. doi: 10.1176/appi.neuropsych.13010013. PMID 25255169